CLINICAL TRIAL: NCT02193737
Title: Effects of Drinking at PACU Discharge After General Anaesthesia With Airway Control on Aspiration, Vomiting and Patients Comfort.
Acronym: I-DRINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I-DRINC
Record Dates: First submitted 2014-05-21; First posted 2014-07-18 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-03

CONDITIONS: Scheduled General Anaesthesia With Airway Control

ARMS (2):
- Early oral fluid recovery. (Experimental)
  Interventions: Procedure: Early oral fluid recovery.
- Delayed oral fluid recovery. (Active Comparator)
  Interventions: Procedure: Delayed oral fluid recovery.

INTERVENTIONS:
Procedure: Early oral fluid recovery.
  Arms: Early oral fluid recovery.
Procedure: Delayed oral fluid recovery.
  Arms: Delayed oral fluid recovery.

SUMMARY:
National guidelines about post-operative fasting after general anesthesia are missing.

Current clinical practices are highly variable and no study has ever evaluated on a large scale the real risk of an early drinks recovery in postoperative period.

The aim of this study is to state the impact of early drinks recovery after general anesthesia with laryngeal mask or endotracheal intubation on the risk of aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgery
* General anaesthesia with laryngeal mask or endotracheal intubation.
* Length of surgery < 4 hours

Exclusion Criteria:

* Emergency surgery
* Intra-cranial, cervical or Ear, Nose and Throat surgery
* Guts surgery with guts anastomosis.
* Glottic topical anesthesia
* Patient with nasogastric tube
* Aspiration during surgery or during PACU stay

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1555 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
To determine if early oral fluid recovery after an elective surgery under general anaesthesia with endotracheal intubation or laryngeal mask increasethe incidence of cough during swallowing, ie aspiration. | 1min
  During first swallowing, patients will be observed to establish if cough occurs during this first swallowing.

SECONDARY OUTCOMES:
To determine if early oral fluid recovery (i.e patient discharged of PACU) after general anaesthesia increases post-operative vomiting during first hour and patient comfort rated on a 10 points scale. | 1 hour
  During a one-hour period after first swallowing, patients will be looked after for any vomiting.
  At the end of day, patients will be asked to rate their postoperative comfort on a 10 points scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Poitiers, Poitiers, Vienne, France